CLINICAL TRIAL: NCT02426983
Title: A Pilot Study Using an NMDA Antagonist to Modulate Transcranial Direct Current Stimulation (tDCS) Effects on Auditory Sensory Memory Processing
Brief Title: Pilot Study Using an NMDA Antagonist to Modulate Transcranial Direct Current Stimulation (tDCS) Effects on Sensory Discrimination
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Dr. Verner Knott, Director, Clinical Neuroelectrophysiology and Cognitive Research Laboratory, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2013008
Record Dates: First submitted 2015-04-13; First posted 2015-04-27 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation; Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Direct Current Stimulation active (Active Comparator): Electrodes will be placed on the scalp overlying the left auditory cortex (anodal electrode) and on the contralateral forehead above the orbit (reference/cathode). Stimulation will be applied using a battery-driven constant-current regulator (Oasis Pro, Edmonton). In active tDCS sessions, the DC current will be initially increased in a ramp-like fashion over 10 s until reaching 2 mA and will be similarly decreased at the end of stimulation. In active tDCS, stimulation will be maintained for a total of 20 minutes. This will occur in two separate sessions, occurring within weeks.
  Interventions: Device: Direct Current Stimulation
- Direct Current Stimulation sham (Sham Comparator): In sham sessions, the device will have the same placement and intensity, but will only be turned on for 30 seconds. The DC current will be initially increased in a ramp-like fashion over 10 s until reaching 2 mA and will be similarly decreased at the end of stimulation. This will occur in two separate sessions, occurring within weeks.
  Interventions: Device: Direct Current Stimulation
- NMDA antagonist active (Active Comparator): Dextromethorphan (DMO), a non-competitive NMDA antagonist, will be delivered in the form of generic Life Brand Clear Cough Syrup DM (Trillium Healthcare Products Inc, Brockville, ON). Each subject will receive a dose of 50 ml DM with no-sugar cranberry juice (100 ml) to drink. This same dose will be delivered in two separate sessions, occurring within weeks.
  Interventions: Drug: Dextromethorphan
- NMDA antagonist placebo (Placebo Comparator): Each subject will receive a dose of a placebo (150 ml of no-sugar cranberry juice) to drink. This same dose will be delivered in two separate sessions, occurring within weeks.
  Interventions: Drug: Dextromethorphan

INTERVENTIONS:
Device: Direct Current Stimulation — Comparison between active Direct Current Stimulation (2 mA, 20 minutes) and Sham stimulation (the device is set up, but only turned on for 30 seconds).
  Conductive saline-soaked rubber electrodes super-imposed on sponge plates will be placed on the scalp overlying the left auditory cortex (anodal electrode) and on the contralateral forehead above the orbit (reference/cathode). Stimulation will be applied using a battery-driven constant-current regulator (Oasis Pro, Edmonton). In active tDCS sessions, the DC current will be initially increased in a ramp-like fashion over 10 s until reaching 2 mA and will be similarly decreased at the end of stimulation. In active tDCS, stimulation will be maintained for a total of 20 minutes. This will occur in two separate sessions, occurring within weeks. For 'sham' stimulation, the device will only be turned on for 30 seconds. This will occur in two separate sessions, occurring within weeks.
  Arms: Direct Current Stimulation active; Direct Current Stimulation sham
Drug: Dextromethorphan — Comparison between Dextromethorphan and a no-sugar placebo. Dextromethorphan (DMO), a non-competitive NMDA antagonist, will be delivered in the form of generic Life Brand Clear Cough Syrup DM (Trillium Healthcare Products Inc, Brockville, ON), which has high dose of DMO (15 mg/5 ml) with no other major additives. Each subject will receive a dose of 50 ml DM with no-sugar cranberry juice (100 ml) to drink from a mug, while wearing a nose plug. This same dose will be delivered in two separate sessions, occurring within weeks. Each subject will receive a dose of a placebo (150 ml of no-sugar cranberry juice) to drink from a mug, while wearing a nose plug. This same dose will be delivered in two separate sessions, occurring within weeks.
  Other Names: Life Brand Clear Cough Syrup DM
  Arms: NMDA antagonist active; NMDA antagonist placebo

SUMMARY:
Transcranial direct current stimulation (tDCS) is a non-invasive form of brain stimulation which uses a very weak constant current to temporarily excite the brain area of interest via small electrodes placed on the scalp. Currently, tDCS is being used as a tool to investigate mental processes (cognition) and motor function (movement) in healthy controls and to treat neurological (i.e. stroke) and psychiatric (i.e. depression and dementia) patients. tDCS has been found to improve motor processes and cognitive performance, including attention and memory functions. This study will attempt to examine the effects of tDCS on a specific aspect of short term memory to sounds measured from electrical activity (EEG) from the top of the scalp. This study will also assess the effect of a drug, dextromethorphan (DMO), commonly found in cough syrup, which is thought to regulate tDCS treatment through brain receptors. The study involves four laboratory test sessions. EEG assessments will be done in two sessions involving 'anodal' tDCS stimulation (to temporarily excite cortical activity locally), one session with DMO treatment and one with placebo treatment, and two sessions involving 'sham' tDCS stimulation (device is turned off), with the same DMO and placebo treatments. These findings will contribute to our understanding of the brain chemistry involved in tDCS treatment and its effects on cognitive abilities.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, medication free
* Non-smoker
* Right-handed

Exclusion Criteria:

* Any current or past Axis I or Axis II disorder including a current or recent history of alcohol/substance abuse
* A clinically significant medical illness or organic brain disorder known to cause psychosis or cognitive impairment
* Any neurological diagnosis (including epilepsy)
* Recent head trauma (<6 months)
* Metallic implants or any electrical device (e.g., pacemaker) in the body
* Major learning disability
* Body mass index >38kg/m¬2
* Use of illicit drugs
* Abnormal hearing

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-09 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
MMN ERP amplitudes as a measure of sensory processing changes | 1 year
  Acute effects of DMO (vs. placebo) and tDCS (vs. sham) on MMN-indexed auditory sensory memory processing
Adverse Events Scores as measure of treatment side effects | 1 year
  Adverse Events and self-reported symptoms after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Impey, Ph.D. (cand.), Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa Institute of Mental Health Research, Ottawa, Ontario, Canada